CLINICAL TRIAL: NCT05989035
Title: Effects of MetAP2 Inhibition on Bioenergetics and Aging-associated Characteristics in Adipose Tissue (BIO-AGE) in Healthy Participants
Brief Title: Effects of MetAP2 Inhibition on Bioenergetics and Aging-associated Characteristics in Adipose Tissue in Healthy Participants
Acronym: BIO-AGE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1389184
Record Dates: First submitted 2023-07-21; First posted 2023-08-14 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Aging
Keywords: adipose tissue; adipocyte

STUDY DESIGN:
Intervention Model Description: This is a prospective single-site study, consisting of two groups of participants. Group 1 will be younger participants between the ages of 18 and 30 years old. Group will be older participants that are 65 years and older. Each participant will have an abdominal subcutaneous adipose tissue (AT) biopsies. Two aliquots from each biopsy will be incubated for conditioned media with and without MetAP2 inhibition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Younger without MetAP2 inhibition (Active Comparator): Participants between 18 and 30 years old without MetAP2 inhibition in conditioned media
  Interventions: Procedure: Abdominal subcutaneous adipose tissue biopsy
- Older without MetAP2 inhibition (Active Comparator): Participants 65 years old and without MetAP2 inhibition in conditioned media
  Interventions: Procedure: Abdominal subcutaneous adipose tissue biopsy
- Younger with MetAP2 inhibition (Experimental): Participants between 18 and 30 years old with MetAP2 inhibition in conditioned media
  Interventions: Procedure: Abdominal subcutaneous adipose tissue biopsy
- Older with MetAP2 inhibition (Experimental): Participants 65 years old with MetAP2 inhibition in conditioned media
  Interventions: Procedure: Abdominal subcutaneous adipose tissue biopsy

INTERVENTIONS:
Procedure: Abdominal subcutaneous adipose tissue biopsy — Fatty tissue biopsy- Participant will be placed in a supine position with arms placed at side while abdominal skin is marked with a skin marker and cleansed with chlorhexidine. Afterwards, the abdominal fatty tissue biopsy will be performed.
  Collect fatty tissue from young and older individuals and gather data on the effect of methionine aminopeptidase protein (MetAP2) inhibition on that fatty tissue in the laboratory.

SUMMARY:
This study is being done to collect Adipose tissue from young and older individuals and gather data on the effect of methionine aminopeptidase protein (MetAP2) inhibition on that Adipose tissue in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1 cohort are male or female participants between 18 and 30 years old
2. Group 2 cohort are male or female participants ≥ 65 years old
3. Body mass index (BMI) ≤ 40 kg/m2
4. Weight stable (±5 kg) for the last 3 months prior to the Screening visit
5. Sedentary (<20 min of activity, 3x/week).
6. Able to speak and understand written and spoken English
7. Willing and able to comply with scheduled visits, laboratory tests, and other study procedures
8. Participant has voluntarily signed and dated an informed consent form, approved by an Institutional Review Board/Independent Ethics Committee, and provided Health Insurance Portability and Accountability Act authorization (HIPAA) or other privacy authorization prior to any participation in study

Exclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus
2. Diagnosis of type 2 diabetes mellitus (HbA1C ≥ 6.5)
3. Insulin use and use of any other medications for diabetes.
4. Use of metformin for polycystic ovarian disease
5. Untreated or poorly controlled hypertension (SBP > 160, DBP > 100)
6. Participants are actively pursuing weight loss and/or lifestyle changes
7. Participants have a sensitivity or allergy to lidocaine
8. Drug or alcohol abuse (> 3 drinks per day) within the last 5 years
9. Any unstable medical condition (i.e., coronary heart disease, stroke, chronic renal failure [serum creatinine should not exceed 1.5-fold the upper laboratory norm and estimated eGFR should not be lower than 60 mL/min/1.73 m2 at screening], chronic hepatic disease, severe pulmonary disease, bleeding disorders, autoimmune disease, active rheumatoid arthritis or other inflammatory rheumatic disorder, or gastrointestinal disease requiring medication)
10. Participants currently taking anti-inflammatory medications within 2 days prior to biopsy or antiplatelet medications within 7 days prior to biopsy, that cannot be safely stopped for study procedures
11. Participants who have a TSH >10 µIU/ml or less than 0.4 µIU/ml
12. Triglycerides >500
13. Pregnant or nursing females or females less than 9 months postpartum.
14. For females only, any new onset (< 3 months on a stable regime) use of oral contraceptives (with the exception of hormone replacement therapy)
15. Tobacco or nicotine containing product use within the past 3 months
16. Major surgery within 4 weeks prior to the Screening Visit
17. Anemia (hemoglobin <11 g/dl in men, <10 g/dl in women) at Screening
18. Participation in studies involving investigational drug(s) within 30 days prior to the Screening Visit
19. Known history of Human Immunodeficiency Virus (HIV), chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C.
20. Any malignancy not considered cured, except basal cell carcinoma and squamous cell carcinoma of the skin (a participant is considered cured if there has been no evidence of cancer recurrence in the previous 5 years)
21. Presence of any condition that, in the opinion of the Investigator, compromises participant safety or data integrity or the participant's ability to complete study visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The effect of MetAP2 inhibition on senescence markers in adipose tissue explants | 4 weeks
  CXCL14 concentration (pg/ml/mg) in conditioned media
The effect of MetAP2 inhibition on adipose tissue quality in adipose tissue explants | 4 weeks
  Adiponectin and resistin concentration (ng/ml/mg) in conditioned media
The effect of MetAP2 inhibition on adipose tissue quality in adipose tissue explants | 4 weeks
  Leptin concentration (pg/ml/mg) in conditioned media

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Sparks, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- AdventHealth Translational Research Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website for AdventHealth Translational Research Institute — https://www.adventhealthresearchinstitute.com/research/translational-research

DOCUMENTS (1):
  • Informed Consent Form (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/35/NCT05989035/ICF_000.pdf